CLINICAL TRIAL: NCT00439673
Title: A Open Label, Phase II, Non Randomized, Clinical Trial of Chemotherapy Treatment With 5-Azacytidine Plus Valproic Acid and Eventually Atra for Patients Diagnosed With Intermediate II and High Risk Myelodysplastic Syndrome (MDS). EudraCT Number 2005-004811-31. GIMEMA Protocol MDS0205
Brief Title: PhII 5-Azacytidine Plus Valproic Acid and Eventually Atra in Intermediate II and High Risk MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS0205
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; 5-Azacytidine; valproic acid; atra; intermediate or high risk; Age ≥18 yearsAge
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Valproic Acid

INTERVENTIONS:
Drug: 5-Azacytidine
Drug: Valproic Acid
Drug: ATRA

SUMMARY:
The primary objective of the trial is to assess the activity of the combined use of Valproic Acid (VPA)in combination with 5-Azacytidine (5-Aza C) in the treatment of MDS.

Activity will be evaluated as percentage of patients achieving complete or partial remission.

DETAILED DESCRIPTION:
Myelodisplastic Syndromes (MDS) are a heterogeneous group of diseases characterized by ineffective hematopoiesis (as a result of increased apoptosis of precursor cells), progressive peripheral cytopenia, with a tendency to evolve to acute leukemia.

The term "syndrome" represents the wide clinical spectrum of this group of diseases, ranging from mild and stable cytopenia, with a low risk of leukemic conversion and a life expectancy of several years, to true pre-leukemia.

The International MDS Risk Analysis Workshop recently developed a consensus risk-based International Prognostic Score System (IPSS) for primary MDS, which has markedly improved prognostic stratification of MDS patients. Following IPSS,it is now possible to identify patients (i.e. Hig-Risk and Intermediate-2-Risk patients) with a bad prognosis (i.e. a life-expectancy < 1 year) due to a high risk of leukemic evolution.

Currently, allogeneic stem cell transplantation represents the only curative therapy for this subgroup of high-risk patients. However, this therapeutic option is often precluded for several reasons (old age, comorbidity, lack of suitable donor).

Among the experimental treatments hitherto tested, 5-Azacitidine (5-Aza) has recently shown promising results. Moreover, the biological experimental data suggest that the association of 5-Aza with histone deacetylase inhibitors, such as Valproic Acid, and with differentiating agents, such as retinoic acid, might be synergistic.

Azacitidine (Aza C), a pyrimidine nucleoside analog, was developed as an antitumor agent. In addition to cytotoxic effects, it induces differentiation of malignant cells in vitro. Aza C inhibits DNA methyltransferase, the enzyme in mammalian cells responsible for methylating newly synthesized DNA, resulting in synthesis of hypomethylated DNA and changes in gene transcription and expression. The mechanism by which Aza C produces its effects is most likely multifactorial. Aza C can produce significant myelosuppression, particularly at higher doses. Aza C could also be acting as a biologic response modifier. The response of hematopoietic progenitors to cytokines is impaired in patients with MDS. This may be attributable in part to abnormalities of the signal transduction pathway downstream from the cytokine receptors. In vitro data suggest that Aza-C can modulate the cytokine signal transduction pathway, rendering sensitive unresponsive cells to the effects of cytokines, partially restoring normal hematopoietic regulation. Incorporation of Aza-C into DNA inhibits DNA methyltransferase and induces DNA hypomethylation. 5-Azacytidine and 5-Aza-2_-deoxycytidine (decitabine), 2 potent inhibitors of cytosine methylation, have shown strong antileukemic activity in acute myeloid leukemia (AML). In addition, both induce trilineage responses in myelodysplastic syndromes (MDS) at dose levels allowing for outpatient management, with moderate myelotoxicity and no significant nonhematologic toxicity.

Azacytidine is the only drug approved by FDA for the treatment of MDS. The median survival for patients with MDS and a Intermediate/high IPSS score, treated with conventional care regimens, is assumed to be 11 months. Patients treated with Azacytidine in the CALGB 9221 trial had a median survival of 18 months. Responses occurred in 60% of patients on the Aza C arm (7% complete response, 16% partial response, 37% improved) compared with 5% (improved) receiving supportive care (P <.001). Median time to leukemic transformation or death was 21 months for Aza C versus 13 months for supportive care (P =.007). Transformation to acute myelogenous leukemia occurred as the first event in 15% of patients on the Aza C arm and in 38% receiving supportive care (P =.001). Furthermore, Aza-C improved quality of life, compared to supportive care.

The opposing actions of histone acetyltransferases (HATs) and histone deacetylases (HDACs) allow gene expression to be exquisitely regulated through chromatin remodelling. Aberrant transcription due to altered expression or mutation of genes that encode HATs, HDACs or their binding partners, is a key event in the onset and progression of cancer. HDAC inhibitors can reactivate gene expression and inhibit the growth and survival of tumour cells. The remarkable tumour specificity of these compounds, and their potency in vitro and in vivo, underscore the potential of HDAC inhibitors as exciting new agents for the treatment of cancer. Histone deacetylase (HDAC) inhibitors have been shown to be potent inducers of growth arrest, differentiation, and/or apoptotic cell death of transformed cells in vitro and in vivo. One class of HDAC inhibitors, hydroxamic acid-based hybrid polar compounds (HPCs), induce differentiation at micromolar or lower concentrations. Studies (x-ray crystallographic) showed that the catalytic site of HDAC has a tubular structure with a zinc atom at its base and that these HDAC inhibitors, such as suberoylanilide hydroxamic acid (SAHA) and trichostatin A, fit into this structure with the hydroxamic moiety of the inhibitor binding to the zinc. HDAC inhibitors cause acetylated histones to accumulate in both tumor and normal tissues, and this accumulation can be used as a marker of the biologic activity of the HDAC inhibitors. Hydroxamic acid-based HPCs act selectively to inhibit tumor cell growth at levels that have little or no toxicity for normal cells. These compounds also act selectively on gene expression, altering the expression of only about 2% of the genes expressed in cultured tumor cells. In general, chromatin fractions enriched in actively transcribed genes are also enriched in highly acetylated core histones, whereas silent genes are associated with nucleosomes with a low level of acetylation. However, HDACs can also acetylate proteins other than histones in nucleosomes. The role that these other targets play in the induction of cell growth arrest, differentiation, and/or apoptotic cell death has not been determined. Our working hypothesis is that inhibition of HDAC activity leads to the modulation of expression of a specific set of genes, which control has been disrupted by ectopic expression of EVI1 or similar oncogene, that, in turn, result in growth arrest, differentiation, and/or apoptotic cell death. The hydroxamic acid-based HPCs are potentially effective agents for cancer therapy and, possibly, cancer chemoprevention.

Valproic acid Valproic acid (VPA, 2-propylpentanoic acid) is an established drug in the long-term therapy of epilepsy. During the past years, it has become evident that VPA is also associated with anti-cancer activity. VPA not only suppresses tumor growth and metastasis, but also induces tumor differentiation in vitro and in vivo. Several modes of action might be relevant for the biological activity of VPA: (1) VPA increases the DNA binding of activating protein-1 (AP-1) transcription factor, and the expression of genes regulated by the extracellular-regulated kinase (ERK)-AP-1 pathway; (2) VPA downregulates protein kinase C (PKC) activity; (3) VPA inhibits glycogen synthase kinase-3beta (GSK-3beta), a negative regulator of the Wnt signaling pathway; (4) VPA activates the peroxisome proliferator-activated receptors PPARgamma and dagger (Rif. 25); (5) VPA blocks HDAC (histone deacetylase), causing hyperacetylation. The findings elucidate an important role of VPA for cancer therapy. VPA might also be useful as low toxicity agent given over long time periods for chemo prevention and/or for control of residual minimal disease. Authors show that the well-tolerated antiepileptic drug valproic acid is a powerful HDAC inhibitor. Valproic acid relieves HDAC-dependent transcriptional repression and causes hyperacetylation of histones in cultured cells and in vivo. Valproic acid inhibits HDAC activity in vitro, most probably by binding to the catalytic center of HDACs. Most importantly, valproic acid induces differentiation of carcinoma cells, transformed hematopoietic progenitor cells and leukemic blasts from acute myeloid leukemia patients. More over, tumor growth and metastasis formation are significantly reduced in animal experiments. Therefore, valproic acid might serve as an effective drug for cancer therapy. These findings constitute a "proof of concept" to use valproic acid for the therapy of acute leukemia and myelodisplastic syndrome.

ATRA

Retinoids have been shown to have a major role in the treatment of APL. There is also in vitro evidence that primary blast cells from FAB groups other than M3 can demonstrate phenotypic evidence of maturation when exposed to retinoid with or without other agents. Additional relevant information on AML/MDS comes from a number of sources:

(I) The addition of retinoid increases the sensitivity of AML blasts to Ara C in vitro.

(II) BCL 2 protein is over-expressed in a proportion of AML cases. There is some evidence that this correlates with treatment response and survival and, since chemotherapy results in apoptotic cell death, this may constitute a mechanism of chemo-resistance. Retinoids down regulate BCL 2 expression AML blasts in vitro. The increased sensitivity of AML blasts to chemotherapy mentioned above, mediated by retinoid, is due to shortening of the BCL 2 half-life.

(III) In a pilot study by Tallman et al, 39 high risk patients with a median age of 65 years, most of whom (n=25) had failed to respond to chemotherapy, were treated with ATRA (150 mg/m2) and LD Ara C. Forty-two percent of patients achieved a CR (25%) or PR (17%) and a further 17% had stable disease.

(IV) In a recent study from M.D. Anderson Cancer Center, Houston, 170 patients with a median age of 66 years with AML or high risk MDS were randomized to receive FAI (fludarabine, Ara C and idarubicin) alone, or FAI combined with either G CSF or ATRA or both. The overall 6 month survival was 49%. In a comparison of ATRA-treated versus ATRA-non-treated patients, there was a more favourable outcome in recipients of retinoids, with CR rates of 56% vs 42% respectively (p=0.06) and superior 6 month survival and event free survival (both p=0.02) but no long-term benefit was demonstrable. In this study the exposure to retinoid was relatively short, namely from day -2 to day +8 of chemotherapy (Rif. 30).

(V) In a recent study from Dusseldorf, 18 patients with MDS and AML secondary to MDS were treated with Valproic Acid (VPA) alone, and 5 patients received a combination of VPA and ATRA. A favourable response was observed in 44% of the patients treated with VPA alone, with a median response duration of 4 (3-9) months. Four of the five patients who subsequently relapsed were treated with VPA + ATRA, two of them responding again. The Authors hypotize that pre-treatment with VPA might be necessary for a synergistic effect of both drugs.

The above evidence suggests that retinoids may be a useful biological response modifier (when combined with chemotherapy and/or VPA) with little or no additional toxicity. Their role will therefore be examined in this trial, in association with 5-Azacytidine and Valproic Acid.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of refractory anemia with excess blasts (RAEB) or refractory anemia with excess blasts in transformation (RAEB-t) according to the French-American-British classification system for MDS with an International Prognostic Scoring System score of INT-2 or High or diagnosis of Myelodysplastic CMMoL per a modified FAB criteria and a relatively high risk of AML transformation;

  * Age ≥18 years;
  * life expectancy ≥3 months;
  * Be unlikely to proceed to bone marrow or stem cell transplantation therapy following remission;
  * Signed written informed consent according to IGH/EU/GCP and national local laws;
  * Eastern Cooperative Oncology Group Performance Status Grade of 0-2 (Appendix D);
  * Serum bilirubin levels ≤1.5 x the upper limit of the normal (ULN) range for the laboratory; higher levels are acceptable if these can be attributed to active hemolysis (as indicated by positive direct Coombs' testing, decreased haptoglobin level, elevated indirect bilirubin and/or lactate dehydrogenase), or ineffective erythropoiesis (as indicated by bone marrow findings);
  * Serum glutamic-oxaloacetic transaminase (aspartate aminotransferase) or serum glutamic-pyruvic transaminase (alanine aminotransferase) levels ≤2 x ULN;
  * Women of childbearing potential may participate, providing they meet the following conditions:
* Must not start a pregnancy throughout the study and for 6 months following the date of the last dose of study medications;
* Must have a negative serum pregnancy test obtained within 48 hours prior to Day 1.

  * Males with female partner of childbearing potential must avoid fathering throughout the study and for 6 months following the date of the last dose of study medication.

Exclusion criteria:

* acute myeloid leukaemia (i.e. bone marrow blasts >30%);
* concurrent malignancy diagnosed in the past 12 months (with the exception of skin basalioma);
* severe renal impairment (creatinine clearance <30 ml/min);
* pregnant or lactating, or are potentially fertile (both males and females) and have not agreed to avoid pregnancy during the trial period;
* they have liver disease characterized by AST and ALT level >2X ULN and total bilirubin > 1.5X ULN (unless due to active hemolysis or ineffective erythropoiesis;
* HIV infection;
* active, uncontrolled HCV or HBV infections or liver cirrhosis;
* clinically relevant neurological diseases;
* psychiatric illness that would prevent granting of informed consent;
* hypersensitivity (known or suspected) to Azacytidine or Mannitol
* prior Treatments: Prior investigational drugs (within 30 days) Radiation therapy, chemotherapy, or cytotoxic therapy for non- MDS conditions within the previous 6 months Growth factors (EPO, G-CSF or GM-CSF) during the previous 21 days Androgenic hormones during the previous 14 days Prior transplantation or cytotoxic therapy, including azacitidine and chemotherapy, administered to treat MDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe LEONE, MD, PHD, Principal Investigator — Università degli studi di Roma La Cattolica
Locations (7):
- Italy (7):
  - USL 8 di Arezzo, Arezzo
  - Azienda Ospedaliera S. G. Moscati, Avellino
  - Università degli studi di Bari, Bari
  - Istituto ematologia e oncologia medica L.A. Seragnoli, Bologna
  - Ospedale Reg. A di Summa, Brindisi
  - Ospedale A. Businco, Cagliari
  - Università degli studi di Roma La Cattolica, Roma

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group
Started | 62
Completed | 26
Not Completed | 36

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 62
Age, Customized [Median (Full Range); unit: years]
  Age | 69.6 [52.9 to 83.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 43
Region of Enrollment [Number; unit: participants]
  Italy | 62

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Trial is to Assess the Efficacy of the Combined Use of Valproic Acid (VPA) in Combination With 5-Azacytidine (5-Aza C) in the Treatment of MDS.
Description: Overall survival
Time Frame: At 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Group
Number analyzed (Participants) | 26
months | 8.3 [3.27 to 21.1]

2. Secondary Outcome: Time to Transformation to AML
Time Frame: At 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Group
Number analyzed (Participants) | 23
months | 53.9 [39.2 to 66.0]

ADVERSE EVENTS:
Time Frame: For 38 months
Description: Non-serious adverse events are not reported.
Groups:
- Study Group: Other adverse events were not included in the final study report, thus, we have included in the present form, all serious adverse events and mortality.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 15/62
Serious Adverse Events (participants affected / at risk) | 24/62
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=62)
Perineal infiltration (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Bronchopneumonic outbreak (Infections and infestations) | 1 (1)
Hemorragic shock (Blood and lymphatic system disorders) | 1 (1)
Right pleuropneumonia (Infections and infestations) | 1 (1)
Local inflamation (General disorders) | 2 (2)
Abscess (General disorders) | 1 (1)
Sepsis (General disorders) | 1 (1)
Sedation (General disorders) | 1 (1)
Fever in neutropenia (General disorders) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Broncopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inflammatory bowel (General disorders) | 1 (1)
Bowel abscess (General disorders) | 1 (1)
Right lung pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperpyrexia and hypoxia (General disorders) | 1 (1)
Confusion and disorientation (General disorders) | 1 (1)
Somnolence and obtundation (General disorders) | 1 (1)
Head and facial contusion (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs of participating centers may disclose their centre's results only after the main study publication has been released, so that a single centre experience can be compared to the study overall results and give a more appropriate view of the study.